CLINICAL TRIAL: NCT06447597
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Phase II/III Clinical Study to Evaluate the Efficacy and Safety of B007 in Subjects With Generalized Myasthenia Gravis
Brief Title: A Clinical Study of B007 in the Treatment of Generalized Myasthenia Gravis.
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai Jiaolian Drug Research and Development Co., Ltd (Industry)
Collaborators: Shanghai Pharmaceuticals Holding Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPH-B007-303
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-06

CONDITIONS: Generalized Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- B007 (Experimental)
  Interventions: Drug: B007
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: B007 — B007 high dose and low dose： Subcutaneous injection was administered on days 1 and 15
  Arms: B007
Drug: Placebo — B007 matched Placebo Subcutaneous injection was administered on days 1 and 15
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of B007 in subjects with generalized myasthenia gravis.

ELIGIBILITY:
Inclusion Criteria:

1. Sign informed consent form;
2. Subjects with generalized myasthenia gravis;
3. Serum AchR(Acetylcholine receptor)-Ab or MUSK-Ab was positive during screening;
4. MG-ADL ≥5 at screening and baseline;
5. Before randomization, subjects received at least one gMG stable dose of SoC, and maintain a stable dose throughout the test;
6. Subjects agree to use effective contraceptive methods for contraception from signing the informed consent form to 1 year after the last dose. Female subjects considered fertile by the investigator must have negative serum pregnancy tests before the first dose.

Exclusion Criteria:

1. Subjects with MGFA I and V type;
2. Subjects usingprescribed drugs;
3. Subjects with a prescribed disease or history of disease;
4. The subjects has prescribed examination abnormalities that are assessed as unsuitable for participation in the study by the investigator;
5. Known history of severe allergic reaction to humanized monoclonal antibodies, or known allergy to any component of B007;
6. Subjects who received live vaccine at the specified time before the first dose and are expected to receive the vaccine at the specified time after the last dose;
7. Subjects who have received major surgery or participated in other clinical trials within the prescribed time before screening;
8. Pregnant and lactating women;
9. Fertile female subjects do not agree to use effective contraception from signing the informed consent form to 1 years after the last dose.
10. Sexually active male subjects who do not intend to use an effective contraceptive method during the trial period or within1 years after the last dose, or male subjects who plan to donate sperm during the trial or within 1 year after the last dose;
11. A history of alcohol or drug abuse within the past 12 months;
12. Other conditions deemed unsuitable for participation in this study by the researchers.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects：MG-ADL（Myasthenia gravis-activities of daily living profile） decreased by ≥2 | Approximately 16 weeks
  Proportion of subjects：MG-ADL decreased by ≥2

SECONDARY OUTCOMES:
Proportion of subjects：subjects without SoC（Standard of Care） change and MG-ADL decreased by ≥2 | Approximately 24 weeks
  Proportion of subjects：subjects without SoC change and MG-ADL decreased by ≥2
Proportion of subjects：subjects without SoC change and QMG(Quantitative Myasthenia Gravis score) decreased by ≥3 | Approximately 24 weeks
  Proportion of subjects：subjects without SoC change and QMG decreased by ≥3
Changes in MGQoL15r (Myasthenia gravis quality of life15-item revised) from baseline. | Approximately 24 weeks
  Changes in MGQoL15r from baseline.
Changes in MGC (Myasthenia gravis composite) from baseline. | Approximately 24 weeks
  Changes in MGC from baseline
Incidence of Treatment-Emergent Adverse Events | Approximately 1 years
  Adverse event type, incidence, duration

CONTACTS AND LOCATIONS:
Locations (18):
- China (18):
  - Peking University First Hospital, Beijing
  - The First Bethune Hospital of Jilin University, Changchun
  - Xiangya Hospital Central South University, Changsha
  - Sichuan Provincial People's Hospital, Chengdu
  - Nanfang Hospital, Southern Medical University, Guangzhou
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou
  - Shandong Provincial Qianfoshan Hospital, Jinan
  - Shandong University Cheeloo College of Medicine, Jinan
  - First People's Hospital of Yunnan Province, Kunming
  - Jiangxi Provincial People's Hospital, Nanchang
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - Shandong University Cheeloo College of Medicine, Qingdao
  - Huashan Hospital, Fudan University, Shanghai
  - Shenzhen Hospital of University of Hong Kong, Shenzhen
  - Renmin Hospital of Wuhan University, Wuhan
  - Tongji Medical College of HUST, Wuhan
  - Tangdu Hospital, Xi'an
  - Affiliated Hospital of Zunyi Medical College, Zunyi